CLINICAL TRIAL: NCT07152977
Title: Description of the Radiological Response of Anoperineal Fistulizing Lesions of Crohn's Disease in Patients Treated With Biotherapy
Brief Title: Description of the Radiological Response of Anoperineal Fistulizing Lesions of Crohn's Disease
Acronym: PéricrohnIRM
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/396/OB; 2018-A03187-48 (Other: ANSM)
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-01

CONDITIONS: Anoperineal Lesions; Crohn's Disease Relapse
Keywords: magnetic resonance imaging; anti-TNF treatment; "Treat-to-target" strategy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Radiological evolution of ano-perineal lesions by MRI — Patients selected retrospectively will have benefited from an MRI at diagnosis and a control MRI during follow-up. They will be selected during a follow-up consultation or a biotherapy injection in a day hospital. Patients selected consecutively are monitored at the Rouen University Hospital for perineal Cohn's disease, treated with Biotherapy: Infliximab, Adalimumab, Ustekinumab, Vedolizumab.

SUMMARY:
The presence of ano-perineal lesions (APL) in Crohn's disease is common and represents a major burden for the patient. More than one-third of patients with Crohn's disease will develop at least one ano-perineal lesion during the course of their disease. The cumulative incidence of APL is approximately 30% at 10 years and 43% at 20 years, regardless of the type of APL.

The appearance of ano-perineal lesions represents an important phase in the progression of Crohn's disease, but they have been little studied to date. There is little consensus regarding their overall management. Indeed, their management is difficult due to their destructive and recurrent nature, and their significant impact on patients' quality of life, continence, and sexuality is significant. The presence of ano-perineal lesions at the time of diagnosis, especially in young patients, is a poor prognostic factor.

DETAILED DESCRIPTION:
Currently, magnetic resonance imaging is the gold standard for diagnosing anoperineal lesions in Crohn's disease. It allows for precise mapping of lesions, and its safety allows for repeated use. MRI is therefore highly effective for diagnosis and can also highlight lesions not identified during clinical examination.

Therapeutic objectives for Crohn's disease are changing, and a new "treat-to-target" strategy is emerging in the guidelines. It consists of closely monitoring clinical symptoms and endoscopic lesions to achieve complete remission. The occurrence of anoperineal lesions has been studied, and relapse is common under anti-TNF alpha therapy. It is conceivable that the treatment of anoperineal lesions could follow the same strategy. However, the role of MRI in monitoring ano-perineal lesions is poorly codified. A Rouen study investigated the feasibility of MRI for the study of ano-perineal lesions and assessed the clinical benefit of anti-TNF treatment in APL due to Crohn's disease, which was associated with a significant improvement in the Van Assche score, particularly T2 hyperintensity, a sign of perineal Crohn's disease activity. The disappearance of contrast enhancement was associated with remission. In 2017, follow-up of these APL patients treated with anti-TNF therapy found twenty-six patients in clinical remission, and 16 of the 26 had a normal MRI, defined by the absence of contrast enhancement or T2 hyperintensity.

The radiological evolution of ano-perineal lesions is also poorly understood. MRI monitoring of anoperineal lesions will be a determining element of the future "Treat-to-target" strategy, in the context of the emergence of new biotherapies and other treatments. Among the anti-TNF agents used in Crohn's disease, only infliximab has been specifically evaluated in anoperineal lesions. (15) Another anti-TNF agent used, adalimumab, has been poorly evaluated.

Data regarding the efficacy of other monoclonal antibodies such as vedolizumab (anti-integrin antibodies) and ustekinumab (anti-IL12 and IL23 antibodies) are currently limited. The main objective of the study is to describe the radiological evolution of patients with Crohn's disease, with fistulizing anoperineal lesion, treated with biotherapy.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients, monitored at the Rouen University Hospital for Crohn's disease, complicated by fistulizing anoperineal lesion, treated with Biotherapy, having benefited from an MRI at the start of treatment and during follow-up.

Exclusion Criteria:

* Minor patients
* Patients with an anoperineal lesion, without Crohn's disease
* Patients who have received surgical treatment with a stoma for perineal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tous les patients majeurs, suivis au CHU de Rouen pour une maladie de Crohn, compliquée de lésion ano-périnéale fistulisante, traités par Biothérapie
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Radiological evolution of patients | at the enrollment visit, at the 1-year visit and at the 3-year visit
  The main objective of the study is to describe the radiological evolution of patients with Crohn's disease, with fistulizing anoperineal lesion, treated with biotherapy. For patients selected retrospectively, they must have had an MRI at the diagnosis of the fistulizing anoperineal lesion and a control MRI during follow-up (at 1 year and at 3 years). The fistulizing ano-perineal lesion is defined radiologically by T2 hyperintensity on the initial MRI.

SECONDARY OUTCOMES:
Clinical course of patients with APL | at the enrollment visit, at the 1-year visit and at the 3-year visit
  Describe the evolution of fecal calprotectin in patients with APL by biological analysis of stools and quantitative data collected
Activity of the fistulizing anoperineal lesion | at the 1-year visit and at the 3-year visit
  Describe the evolution of the activity score of the fistulizing anoperineal lesion by the PDAI score. The PDAI Score is collected during follow-up, at 1 year in patients treated with biotherapy: it focuses on 5 items: type of lesion, degree of induration, discharge, sexual impact and pain; each item is subdivided into 5 severity scores ranging from 0 to 4.
Factors associated with radiological response | at the 1-year visit and at the 3-year visit
  Describe the factors associated with radiological response by assessment of the use of surgical management

CONTACTS AND LOCATIONS:
Locations (1):
- University Rouen Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.